CLINICAL TRIAL: NCT05480631
Title: COMPARATIVE ANALYSIS OF INNOVATIVE BONE HEALING TECHNIQUES IN MANDIBLE BONE DEFECTS
Brief Title: COMPARATIVE ANALYSIS OF INNOVATIVE BONE HEALING TECHNIQUES
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Samreen Malik, Doctor (MDS trainee), Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-1835/DUHS/approval/2020
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: To Assess the Bone Healing in Fracture Mandible Defects
Keywords: Concentrated growth factor, bone density, mandible fracture
MeSH Terms: conditions — Mandibular Fractures | interventions — Transplantation, Autologous; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): group A- autograft
  Interventions: Procedure: autograft
- group B (Experimental): group B- concentrated growth factor with autograft
  Interventions: Procedure: autograft with addition of concenterated growth factor
- Group C (Experimental): group C- concentrated growth factor with xenograft
  Interventions: Procedure: xenograft with concentrated growth factor

INTERVENTIONS:
Procedure: autograft — autologous bone placed in the defect and then be secured with mini-screws to fill the fracture defect gap
  Arms: Group A
Procedure: autograft with addition of concenterated growth factor — the bone particulate harvested from the donor site will then be mixed with concentrated growth factor to bridge the fracture defect.
  Arms: group B
Procedure: xenograft with concentrated growth factor — xenogenic bovine bone particulate mixed with platelet-derived concentrated growth factor to be held in place of fracture defect site.
  Arms: Group C

SUMMARY:
the study intends to observe the outcome of interventions (concentrated growth factor with autograft and xenograft) used to expedite bone healing and adaptation with minimal side effects. Three different modalities are being used to bridge the mandibular fracture defects (>5mm-<5cm). Those modalities include group A- autograft, group B-autograft with concentrated growth factor, and group C- xenograft with concentrated growth factor. the outcomes are measured in terms of acquired bone density (Hounsfield unit) that is obtained at the 4th and 6th month post-operatively via cone-beam computed tomography.

DETAILED DESCRIPTION:
Study Design:

Randomized clinical trial

Study Population:

The study will be conducted on patients with mandible fracture defects, exclusively of defect sizes ranging from 5mm to 5cm.

Study Settings:

Department of Oral and Maxillofacial Surgery of

* Dr.Ruth K.M PFAU/ Civil Hospital Karachi
* Ojha Hospital and associated Out Patient Departments. The study will be conducted on patients with mandible fracture defects, exclusively of defect sizes ranging from 5mm to 5cm.

Sampling Technique:

• Non-probability purposive sampling was done in participants fulfilling the inclusion criteria of the study. The diagnosis was made by evaluation of pre-operative Orthopantamamogram along with clinical examination. The defect of the fractured bone was measured from Orthopantomagram then the patient's general physical examination and detailed history were taken. Written and verbal consent was taken by informing the patient regarding all the possible favorable and unfavorable outcomes of the study. Once the consent was taken, Proforma was filled by the principal investigator followed by randomization. Participants in then allocated to any of the three groups that were disclosed via envelope. A total of 60 envelopes were made in three groups that are 20 out of which were of group A receiving autograft as a reconstruction option. Other 20 envelopes were of group B receiving autograft with concentrated growth factor whilst 20 envelopes were of group C receiving xenograft with concentrated growth factor. Participants were asked to randomly pick any of the envelope disclosing the group they were allocated to.

Sample Size A total of 60 subjects were recruited and divided into 3 groups, 20 subjects in each group sample size was calculated using open epi online software.

3.6 Study Duration 2 years after synopsis approval. Inclusion Criteria

* Aged 18-40
* Male/female
* Mandible fracture (symphysis, parasymphysis, and body)
* Defect gap of bone >5mm and <5cm.
* Non-union fracture. (Fracture that does not heal after 8 weeks of treatment is known as a non-union)
* Mal-union (when the fracture segments are not in anatomical alignment and heals in that way forming a bone between displaced segments)
* Delayed union (Fracture which takes greater than 5 weeks to repair is a delayed union) Exclusion Criteria
* Systemic disease involvement such as diabetes mellitus.
* Bone-related disorders such as osteoarthritis,
* Undergoing Chemo and or radiotherapy
* Gunshot trauma with more than 5cm bone defect
* Fracture with open wounds Study Parameters Study Variables
* Bone healing
* Concentrated Growth Factor
* Autograft
* Bovine xenograft Outcome Variables
* Bone healing (bone density) Exposure Variables
* Concentrated Growth Factor
* Autograft
* Bovine xenograft

Ethical Considerations:

Patient's voluntary participation was ensured for this study with their informed verbal and written consent. The information was kept confidential. Only the authorized principal and/or co-investigators were allowed to access the patient's data. Patients were allowed to withdraw from the study at any given point and were also provided with the contact information of concerned authorities in case of communicating their issues regarding the study.

Ethical approval for the study was taken from DUHS reference number: Institutional Review Board-1835/Approval/2020

Data Collection Procedure:

Once the definitive diagnosis is made and the participant is recruited to the allocated group after randomization, consent is taken and the participant's detailed history Proforma is filled. Then the fracture is assessed over a radiograph OPG (Orthopantomogram) categorizing it into either malunion, non-union, or delayed union.

Preparation of concentrated growth factor:

concentrated growth factor was prepared in a centrifuge machine by following standard protocol, machine that was used was product name: Benchtop PRP, PRF, concentrated growth factor, and serial no XX2201XF008. The autologous blood of around 10cc was taken in an empty red top vacutainer tube and is directly placed in a centrifuge machine with a contralateral tube filled with water for balancing purposes. The drawn blood was immediately transferred to a centrifuge machine to avoid clotting. The pre-setting concentrated growth factor option was selected that has an acceleration cycle of 30 sec followed by 2min revolutions at 2700rpm, then followed by 4min of revolutions at 2400rpm, then 4min at 2700rpm leading to 3 min at 3000rpm, and after which the deceleration phase started that lasts for 36 seconds.

Surgical procedure:

After taking Anesthesia Administration Assembly measures, under general anesthesia opting for adequate exposure and scrubbing was undertaken. Local anesthesia containing xylocaine 2% with adrenaline 1:200,000, was injected in the buccal sulcus of the site of fracture. An intra-oral vestibular incision was then given to raise a full-thickness flap in order to expose the fracture adequately; the mental nerve is located and secured alongside bleeding is controlled to assess the fracture site. After removing granulation tissue and mal-aligned bony fragments (in case of mal-union fracture) the size of the defect was gauged using a millimeter scale. Occlusion is restored and bony fragments are held in the best possible anatomic location. Titanium mini-plates are held in place for fixation of fracture whilst the defect is restored and filled with either autograft, autograft with concentrated growth factor, or bovine xenograft with concentrated growth factor. Once the graft is stabilized soft tissue is re-approximated using Vicryl 3.0 sutures.

Surgical procedure for harvesting autograft from intraoral site In cases where autograft was intended to utilize, a pre-operative evaluation was done via assessing the radiograph and palpation. The inferior alveolar nerve block was given then the incision was given at the buccal site just medial to the external oblique ridge from there the extension of the incision is made towards the retromolar pad area. The incision ascending towards Ramal height was kept at the level of the occlusal plane of the mandibular second molar tooth to avoid exposure to the buccal fat pad or injury to the buccal artery. A full-thickness flap was raised above the external oblique ridge and osteotomy was done following 1/3rd thickness from the buccal cortical aspect of the ramus. The desired chunk of not more than 1cm was taken. Osteotomy cuts are inferior ramus cut, and superior ramus cut whilst anterior body cut and inferior to external oblique ridge cut was made with a bur. The anterior cut was kept behind the body and the superior cut was kept below the level of the coronoid, however, this site can provide up to 40mm long grafts but the required donor site defect was not more than 9mm maximum in all groups. Conventionally ramus can provide up to half of its thickness graft in situations where the only graft is intended whilst this study took only 1/3 of the thickness as per requirement. The harvested bone in group "A" participants is kept in place in the defect and secured with mini-screws.

Mechanical Mixing Of concentrated growth facto with Bone Particulates The autologous bone is crushed and mixed with concentrated growth facto via mechanical means similarly, bone particulate of Xeno-graft are also integrated with concentrated growth facto to form a consistent pliable buffy tissue that can be manipulated according to defect size.

Evaluation over Cone Beam Computed Tomography:

Post-operatively Cone Beam Computed Tomography was conducted in all patients in the 4th and 6th months; the machine used was of brand Ville system medical model Uni-Tech Scientific series 16020502. The Cone Beam Computed Tomography for evaluation and tabulation of Bone Mineral Density from the region of interest that is occlusal to the fracture defect was done by assessing the grey level on Cone Beam Computed Tomography by a radiology specialist

ELIGIBILITY:
Inclusion Criteria:

* Male/female
* Mandible fracture (symphysis, parasymphysis, and body)
* Defect gap of bone >5mm and <5cm.
* Non-union fracture. (Fracture that does not heal after 8 weeks of treatment is known as a non-union)
* Mal-union (when the fracture segments are not in anatomical alignment and heals in that way forming a bone between displaced segments)
* Delayed union (Fracture which takes greater than 5 weeks to repair is a delayed union)

Exclusion Criteria:

* Systemic disease involvement such as diabetes mellitus.
* Bone-related disorders such as osteoarthritis,
* Undergoing Chemo and or radiotherapy
* Gunshot trauma with more than 5cm bone defect
* Fracture with open wounds

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
bone density | 6 months
  acquired bone density in region of interest via cone beam computed tomography expressed in Hounsfield units

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of health sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No